CLINICAL TRIAL: NCT03574532
Title: A Retrospective Non-Interventional Study to Determine the Epidemiology and Evaluate the Burden of Disease in Respiratory Syncytial Virus/Human Metapneumovirus and Influenza A Infected Hospitalized Patients (Adults and Children) at Selected European Sites
Brief Title: A Study to Determine the Epidemiology and Evaluate the Burden of Disease in Respiratory Syncytial Virus/Human Metapneumovirus and Influenza A Infected Hospitalized Participants (Adults and Children)
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108444; NOPRODRSV4001 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospitalized adults with RSV, hMPV and influenza A infections: Respiratory Syncytial Virus (RSV)/Human Metapneumovirus (hMPV) and Influenza A Infected adults that required hospitalization or were infected by these viruses while being hospitalized during the prespecified recent past season(s) will be retrospectively observed to describe the proportion and burden of the different types of respiratory pathogens. The primary data source for this study will be the medical records of each participating participant.
- Hospitalized infants/children with RSV or hMPV infection: Respiratory Syncytial Virus (RSV)/Human Metapneumovirus (hMPV) and Infected Infants/Children that required hospitalization or were infected by these viruses while being hospitalized during the prespecified recent past season(s) will be retrospectively observed to describe the proportion and burden of the different types of respiratory pathogens. The primary data source for this study will be the medical records of each participating participant.

SUMMARY:
The purpose of this study is to describe the clinical and economic burden in adults and infants/children less than or equal to 5 years of age by type of respiratory pathogen (respiratory syncytial virus [RSV], influenza A, and human metapneumovirus [hMPV] in adults; RSV and hMPV in infants/children) based on medical resource utilization; rate and type of complications during and after hospitalization; mortality; rate and reasons of re-hospitalization related to index hospitalization; post-discharge care information and International Classification of Diseases 9th/10th revision (ICD-9/10)/Diagnostic-related Group (DRG) codes used (distribution).

ELIGIBILITY:
Inclusion Criteria:

* Adult greater than or equal to (>=) 18 years of age or infant/child less than or equal to (=<) 5 years of age
* Participants hospitalized must have documentation of a confirmed diagnosis by PCR during the prespecified recent past season(s): RSV, influenza A, or hMPV infection in adults RSV or hMPV in infants/children (The first hospitalization in the season of data collection with confirmed diagnosis by PCR is considered the index hospitalization)
* Participants may include those hospitalized in the season of data collection with or without symptoms of a respiratory viral infection (including those of nosocomial origin), and/or to treat complications of viral infections, including patients admitted to the intensive care unit (ICU)
* Hospitalized greater than (>) 24 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population consists of participants hospitalized and had a polymerase chain reaction (PCR) confirmed respiratory infection; respiratory syncytial virus [RSV], influenza A, and human metapneumovirus [hMPV] in adults; RSV or hMPV in infants/children).
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Burden as Measured by Medical Resource Utilization, Complications, Mortality, Re-hospitalizations and Post Discharge Care Information | Up to 6 months after discharge
  Number of participants with medical resource utilization, complications, mortality, re-hospitalizations and post discharge care information will be assessed.

SECONDARY OUTCOMES:
Number of Participants (Adults) with RSV, Influenza A and hMPV Infections | During hospitalization (up to maximum 12 months)
  Number of Adult participants with RSV, Influenza A and hMPV Infections will be reported.
Number of Participants (infants/children) with RSV and hMPV Infection | During hospitalization (up to maximum 12 months)
  Number of infants/children participants with RSV and hMPV infection will be reported.
Number of Participants in Various Subgroups of Hospitalized Patients by Type of Respiratory Pathogen | During hospitalization (up to maximum 12 months)
  Number of participants in various subgroups (eg, comorbidities, premature infants, elderly, immunocompromised) of Hospitalized Patients by Type of Respiratory Pathogen (RSV, influenza A, and hMPV in adults and RSV and hMPV in infants/children less then or equal to (<=) 5 years of age) will be characterized.
Symptoms of Participants Presenting at Hospital | At admission (Day 1) and at discharge
  Symptoms of Participants Presenting at Hospital (outpatient clinic, emergency room/emergency department [ER/ED], or general ward) and at discharge will be assessed.
Number of Participants Without Presenting Symptoms of Acute Respiratory Tract Infection (ARTI) | During hospitalization (up to maximum 12 months)
  Number of participants without presenting symptoms among participants with PCR-confirmed RSV, influenza A, or hMPV infections of ARTI will be reported.
Number of Participants with Respiratory Infections of Nosocomial Origin With or Without Presenting Symptoms | During hospitalization (up to maximum 12 months)
  Number of participants with respiratory infections of nosocomial origin with or without presenting symptoms among participants with PCR-confirmed RSV, influenza A, or hMPV infections will be reported.
Patient Journey | During hospitalization and up to 6 months after discharge
  The number of patients admitted to different hospital-locations (ED/ER department, Ward, Outpatient clinic, ICU, Other), their provenances, the number of patients being transferred to ICU and the number of patients being thereafter re-hospitalized will be assessed.
Criteria Applied for the Index-Hospitalization, Transfer to ICU, Discharge From Hospital | At admission, at ICU admission, at discharge (up to maximum 12 months)
  The distribution of the primary reasons for the index-hospitalization, the distribution of the primary reasons for ICU transfer, the distribution of the criteria used to discharge from the index-hospitalization (including hospital recovery scale (HRS) and oxygen saturation) will be assessed.
Participant's Clinical Status Assessed by Hospital Recovery Scale (HRS) | Baseline, Day 4, Day 6 and Day 14
  The hospital recovery scale assesses a participant's clinical status. The scale provides 6 mutually exclusive conditions ordered from best to worst: 1) not hospitalized; 2) non-ICU hospitalization, not requiring supplemental oxygen; 3) non-ICU hospitalization, requiring supplemental oxygen; 4) admitted to the ICU, not requiring invasive mechanical ventilation; 5) requiring invasive mechanical ventilation; and 6) death.
Change of National Early Warning Score (NEWS) for Adults at Admission, Day 3, and Day 6 | At admission (Day 1), Day 3, and Day 6
  The NEWS provides guidance for 3 scores: Low score (1-4) should prompt assessment by a competent registered nurse who should decide if a change to frequency of clinical monitoring or an escalation of clinical care is required; Medium score (5-6) should prompt an urgent review by a clinician skilled with competencies in the assessment of acute illness; and High score (7 or more) should prompt emergency assessment by a clinical team/critical care outreach team with critical-care competencies.
CRB-65 Scoring System at Admission to the Hospital for Adults with Lung Disease and the Relevance on Medical Resource Utilization (MRU) by type of Respiratory Pathogen | At admission (Day 1)
  Confusion, respiratory rate greater than or equal to (>=) 30/minute, low systolic less than (<) 90 millimeter of mercury (mm Hg) or diastolic less than or equal to (=<) 60 mm Hg blood pressure, age >= 65 years (CRB-65) scoring system at admission to the hospital for adults with lung disease and the relevance on MRU by type of Respiratory Pathogen will be assessed. CRB-65 Scale ranges from 0 to 4. Score 0 = Very low risk of death, Score 1 and 2 = Increased risk of death and 3 or 4 = High risk of death.
Acute Physiologic and Chronic Health Evaluation (APACHE II) Scores in Adults at ICU Admission and the Relevance on MRU by Type of Respiratory Pathogen | At ICU admission (up to maximum 12 months)
  The APACHE II is a validated severity of disease classification system. It uses a point score based on initial values of 12 routine physiologic measurements (temperature, mean arterial pressure, heart rate, respiratory rate, oxygenation, arterial pH, serum sodium, potassium, and creatinine, hematocrit, white blood cell count, Glasgow coma score), age, and previous health status to provide a general measure of severity of disease. An increasing score (range 0 to 71) is closely correlated with subsequent risk of hospital death for intensive care admissions.
Simplified Acute Physiology Scores 3 (SAPS 3) in Adults at ICU Admission and the Relevance on MRU by Type of Respiratory Pathogen | At ICU admission (up to maximum 12 months)
  The SAPS 3 consists of 20 variables: age, co-morbidities, use of vasoactive drugs before ICU admission, intrahospital location before ICU admission, and length of stay in the hospital before ICU admission, reason(s) for ICU admission, planned/unplanned ICU admission, surgical status at ICU admission, anatomic site of surgery, and presence of infection at ICU admission and place acquired, lowest estimated Glasgow coma scale, highest heart rate, lowest systolic blood pressure, highest bilirubin, highest body temperature, highest creatinine, highest leukocytes, lowest platelets, lowest hydrogen ion concentration (pH), and ventilatory support and oxygenation. Score varies from a minimum of 0 points to a maximum of 217 points. Higher scores indicate higher severity.
Medical Resources Utilization by Type of Virus Infection | Baseline
  MRU in adults by type of virus infection (RSV A, RSV B, influenza A, influenza B, hMPV, any other virus infection if available) at baseline that is before hospitalization will be collected.
Medical Resources Utilization by Estimated Glomerular Filtration Rate (eGFR) | Baseline
  MRU in adults by eGFR at baseline that is before hospitalization will be collected. The glomerular filtration rate is an indicator of renal function and is calculated based on serum creatinine.
ReSVinet score used at Time of Admission to the Hospital in Infants/Children, and Relevance on MRU by Type of Respiratory Pathogen | At Admission (Day 1)
  ReSVinet scale is based on seven parameters (feeding intolerance, medical intervention, respiratory difficulty, respiratory frequency, apnoea, general condition, fever) which are assigned different values (from 0 to 3) for a total of 20 points. Higher scores indicate higher severity.
Levels of White Blood cell During Hospitalization | During hospitalization (up to maximum 12 months)
  Levels of White Blood cell Count during hospitalization will be reported.
Levels of Neutrophils During Hospitalization | During hospitalization (up to maximum 12 months)
  Levels of Neutrophils during hospitalization will be reported.
Levels of Procalcitonin During Hospitalization | During hospitalization (up to maximum 12 months)
  Levels of Procalcitonin during hospitalization will be reported.
Levels of C-Reactive Protein During Hospitalization | During hospitalization (up to maximum 12 months)
  Levels of C-Reactive Protein during hospitalization will be reported.
Levels of Viral Load During Hospitalization | During hospitalization (up to maximum 12 months)
  Levels of Viral Load during hospitalization will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (2):
- Universitätsklinikum Würzburg, Würzburg, Germany
- Hosp. Univ. de La Princesa, Madrid, Spain